CLINICAL TRIAL: NCT05692401
Title: Weight Change With Controlled Ankle Movement (CAM) Boot Use
Acronym: CAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study recruitment stopped due to recruitment problems
Sponsor: Nell Blake, DPM (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor-Investigator, Nell Blake, DPM, Assistant Profesor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY 00021093
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Ankle Injuries; Foot Injuries and Disorders; Body Weight Changes
Keywords: controlled ankle movement; CAM boot
MeSH Terms: conditions — Ankle Injuries; Foot Injuries; Disease; Body Weight Changes | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): CAM boot prescribed as standard of care. No nutritional guidelines or upper body exercises instructions provided. Height and weight recorded at enrollment and final visit.
- Nutrition and Exercise Instruction (Active Comparator): CAM prescribed as standard of care. Nutritional guidelines provided and upper body exercise instructions provided. Height and weight recorded at enrollment and final visit. Subjects in this group will undergo a follow up interview that will ultimately be used to examine and assess the helpfulness of the intervention in preventing weight for CAM boot wearing patients.
  Interventions: Behavioral: Nutrition and Exercise Instruction

INTERVENTIONS:
Behavioral: Nutrition and Exercise Instruction — Eating and exercise patterns. Educational handouts and instructions will be provided, which are intended as a guide for subjects in intervention group. Subjects will also be given a Patient Diary to complete their daily meal intake and physical exercises. Use of and return of the diary is optional but encouraged. It has been found that use of a patient diary to record food intake keeps one from eating more than they planned and can be a useful tool in weight control.
  Arms: Nutrition and Exercise Instruction

SUMMARY:
The purpose of the study is to determine if patients wearing a CAM boot have a change in weight compared to patients who wear a CAM boot and are provided nutritional guidelines and perform upper body exercises.

DETAILED DESCRIPTION:
The study objectives include: 1) Determine if patients wearing a CAM (Controlled Ankle Movement) boot have a change in weight compared to patients who wear a CAM boot and are provided nutritional guidelines at the time the CAM is dispensed and perform upper body exercises through the treatment period. 2) Determine, if weight is gained or lost, the average amount gained/lost over the treatment period. 3) To qualitatively explore if the intervention helped to prevent gain weight during post-operative recovery when CAM boot is used

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years
* Participants with foot or ankle injury who are prescribed a CAM boot as standard of care
* Participants willing to have height and weight measured at the time of enrollment and final visit
* Participant is able to provide voluntary, written consent
* Fluent in written and spoken English
* Participant in the opinion of the Principal Investigator, is able to understand the clinical investigation

Exclusion Criteria:

* Age less than 18 years
* Pregnant women
* Participants with vertigo or other balance issues
* Participants unable to provide informed consent
* Participants with foot or ankle injury who will not be wearing a CAM boot
* Participants unable/unwilling to perform upper body exercises and follow nutrition recommendations

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Weight change | 12 weeks
  Height and weight recorded at enrollment and discontinuation of CAM boot

CONTACTS AND LOCATIONS:
Overall Officials: Nell Blake, DPM, Principal Investigator — Penn State Health Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No